CLINICAL TRIAL: NCT00745433
Title: REPAMET 2: Observational Study of the Switch From Metformin Monotherapy to Bitherapy With Metformin and Repaglinide
Brief Title: Switch From Metformin Monotherapy to a Bitherapy With Metformin and Repaglinide
Acronym: REPAMET 2
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: AGEE-3558
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Repaglinide add-on to metformin.
  Interventions: Drug: repaglinide; Drug: metformin

INTERVENTIONS:
Drug: repaglinide — Start dose and frequency at the discretion of the physician following clinical practice
  Other Names: NovoNorm®
Drug: metformin — Start dose and frequency at the discretion of the physician following clinical practice

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to investigate the efficacy (e.g. glycemic control) and safety (e.g. hypoglycemic episodes) when adding repaglinide to a monotherapy of metformin in type 2 diabetic patients under normal clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Metformin monotreatment
* HbA1c greater than 7%
* Treatment according to SPC
* Informed consent obtained

Exclusion Criteria:

* Any contraindication to the use of repaglinide (according to the SPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any subject with type 2 diabetes treated with metformin
Sampling Method: Non-Probability Sample
Enrollment: 906 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | After 12-20 weeks.

SECONDARY OUTCOMES:
PPG | After 12-20 weeks.
Number of hypoglycemic events | After 12-20 weeks.
Variability in FPG (Fasting Plasma Glucose) | After 12-20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Brussels, Belgium

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com